CLINICAL TRIAL: NCT06009731
Title: DIAPHRAGMATIC SPECKLE TRACKING DURING SPONTANEOUS BREATHING TRIAL
Acronym: DIAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2023_843_0040
Record Dates: First submitted 2023-07-18; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-07

CONDITIONS: Weaning; Spontaneous Breathing Trial; Mechanical Ventilation; Speckle Tracking; Strains; Diaphragm
Keywords: weaning; spontaneous breathing trial; mechanical ventilation; speckle tracking; Strains; diaphragm
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients undergoing mechanical ventilation

SUMMARY:
Currently, measurement of transdiaphragmatic pressure (Pdi) using oesophageal and gastric balloons is the gold standard for the assessment of diaphragmatic effort. This technique is relatively invasive and its interpretation may be complex. The diaphragmatic longitudinal strain (LSdi) and strain rate (LSRdi) might provide additional information in the assessment of diaphragmatic effort and movement during SBT, allowing early detection of diaphragmatic dysfunction. Patients will be monitored during a 30-120 minutes SBT consisting of no assistance on the ventilator using CPAP with a pressure level of 0 cmH2O. Parameters to evaluate diaphragm function will include diaphragmatic strain (LSdi and LSRdi), diaphragmatic thickening fraction (TFdi), and airway occlusion pressure (ΔP0.1 and ΔPocc). These parameters will be measured immediately before ('baseline') the SBT, as well as 2 minutes ('early' assessment), 15 ('intermediate' assessment) and 30 minutes ('late' assessment) after the beginning of the SBT.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients (≥18 years old) undergoing mechanical ventilation for at least 24h (regardless of the reason of intubation)
* patients fulfilling criteria for an SBT
* patients will have to be able to trigger ventilator breaths with a reasonable level of assistance,
* patients with lack of severe impairment in gas exchange,
* patients that not require significant hemodynamic support.
* Patients will be recruited by the study coordinator following completion of informed consent from the patient or legally authorized substitute decision maker.

Exclusion Criteria:

* Use of pressure support during the SBT.
* Severe hemodynamic instability (>30% increase in vasopressors in the last 6 hours or norepinephrine > 0.5 µg/kg/min).
* Severe or very severe chronic obstructive pulmonary disease (COPD) according to the GOLD criteria (stage III: FEV1 30-50% predicted; stage IV: FEV1 < 30% predicted).
* Known or suspected severe or progressive neuromuscular disorder likely to result in prolonged or chronic ventilator dependence
* Clinical judgement of the attending physician.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients (≥18 years old) undergoing mechanical ventilation for at least 24h (regardless of the reason of intubation) and fulfilling criteria for an SBT will be included in the study. Briefly, to be eligible for an SBT, patients will have to (i) be able to trigger ventilator breaths with a reasonable level of assistance, (ii) lack of severe impairment in gas exchange, and (iii) not require significant hemodynamic support. Patients will be recruited by the study coordinator following completion of informed consent from the patient or legally authorized substitute decision maker.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
changes of diaphragmatic longitudinal strain between baseline and during Spontaneous breathing trial | 7 days
  diaphragmatic longitudinal strain is LSdi Spontaneous breathing trial is SBT
changes of diaphragmatic longitudinal strain strain rate between baseline and during Spontaneous breathing trial | 7 days
  diaphragmatic longitudinal strain strain rate is LSRdi Spontaneous breathing trial is SBT

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No